CLINICAL TRIAL: NCT03425136
Title: Scaling up the Systems Analysis and Improvement Approach for Prevention of Mother-to-Child HIV Transmission in Mozambique
Brief Title: Systems Analysis and Improvement Approach for Prevention of MTC HIV Transmission
Acronym: SAIA-SCALE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Ministry of Health, Mozambique (Other Government); Health Alliance International (Other); Fred Hutchinson Cancer Center (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kenneth Sherr, Study Principal Investigator, University of Washington
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000645; 1R01MH113435 (NIH)
Record Dates: First submitted 2018-01-26; First posted 2018-02-07 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: HIV
Keywords: Prevention of Mother-to-Child HIV Transmission; HIV; PMTCT

STUDY DESIGN:
Intervention Model Description: A three-wave stepped-wedge (phased-in) cluster randomized trial, with districts as the unit of randomization (and outcomes assessed at the clinic/individual level within each district)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAIA (Systems Analysis & Improvement) (Experimental): Intervention is a five-step package of industrial engineering methods known as SAIA (the systems analysis and improvement approach) delivered by district maternal and child health managers to subordinate health facilities that provide prevention of mother-to-child HIV services.
  Interventions: Other: Systems Analysis and Improvement Approach (SAIA)
- Control (No Intervention): Routine provision of prevention of mother-to-child HIV transmission services and routine support from district maternal and child health managers to subordinate facilities.

INTERVENTIONS:
Other: Systems Analysis and Improvement Approach (SAIA) — Five-step systems analysis and iterative improvement cycles applied by district maternal and child health supervisors to subordinate health facilities providing prevention of mother-to-child HIV transmission services at the facility level.
  Arms: SAIA (Systems Analysis & Improvement)

SUMMARY:
Optimizing the prevention of mother-to-child HIV transmission cascade minimizes drop offs from one step to the next to maximize the benefits of antiretroviral therapy on maternal health and pediatric survival, growth, and development. This proposal scales-up a health systems intervention (the systems analysis and improvement approach - SAIA) that packages systems engineering methods (including cascade analysis, flow mapping, and continuous quality improvement) and was previously shown to be effective in improving the prevention of mother-to-child HIV transmission cascade. By spreading the SAIA through routine district management structures, and studying the implementation process, this study will build evidence on how to achieve rapid, sustainable and scalable improvements in services that can dramatically improve population health in resource limited countries.

DETAILED DESCRIPTION:
Despite significant increases in global health investment and the availability of low-cost, efficacious interventions designed to prevent mother to child HIV transmission (PMTCT) in low and middle income countries with high HIV burden, the translation of these scientific advances into effective delivery strategies has been slow, uneven and incomplete. As a result, pediatric HIV infection remains largely uncontrolled. The introduction of the Option B+ strategy - where HIV-infected pregnant women rapidly initiate lifelong antiretroviral therapy (ART) independent of disease status - has the potential to dramatically reduce HIV transmission during pregnancy, birth and the breastfeeding period, and as a result, it has been scaled up throughout high HIV burden countries in sub-Saharan Africa. Despite these significant investments to scale-up Option B+, results have been poor, with high rates of loss to follow-up and low viral suppression, leading to continued HIV transmission to children and HIV-associated morbidity among mothers. A previous research project (the Systems Analysis and Improvement Approach - or SAIA - cluster randomized trial) demonstrated that a package of systems engineering tools including cascade analysis, process mapping, and continuous quality improvement, was effective at improving flow through the PMTCT cascade across three sub-Saharan African countries. The overall goal of this application is to develop a model to deliver the SAIA intervention (SAIA-SCALE) that is led by district maternal and child health (MCH) supervisors (rather than research nurses), to serve as a foundation for national scale-up. We propose to implement the SAIA intervention in all districts in one province in Mozambique using MCH supervisors as disseminating agents, who will implement SAIA in subordinate health facilities. Using a three-year phased-in design, 12 districts will be randomly allocated into three implementation waves, and a mixed-methods evaluation will be used to assess the impact of the intervention. Our specific aims are to: Aim 1: Develop an effective district-based dissemination and implementation strategy for the SAIA intervention (SAIA-SCALE), using the RE-AIM model to evaluate the program's Reach, Effectiveness, Adoption, Implementation, and Maintenance; and Aim 2: Using activity based micro-costing and mathematical models of HIV transmission, estimate the budget and program impact from the payer perspective to scale-up the SAIA intervention compared to the standard of care. The results of this implementation research are expected to generate knowledge of global health significance, and by providing a real-world implementation model for the SAIA intervention and programmatically relevant information, is designed to lead to rapid policy translation for future scale-up in countries with high burden of HIV and weak PMTCT delivery systems.

ELIGIBILITY:
Inclusion Criteria • Woman/infant pair attending pMTCT and linked pediatric HIV screening and treatment services at a public sector health facility

Exclusion Criteria

• None

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Maternal retention in care, evaluated using clinic registry data | 6-months post ART initiation
  Women retained in care (picked up their 6-month pharmacy refill within 15 days of scheduled pickup)

SECONDARY OUTCOMES:
Maternal viral load assessment, evaluated using clinic registry data | Within 1 month of delivery (birth)
  Proportion of women on ART with viral load assessment
Early Infant Diagnosis for HIV, evaluated using clinic registry data | within 8 weeks of birth
  Proportion of HIV-exposed infants tested for HIV (PCR) within 8 weeks of birth
Facility Delivery, evaluated using clinic registry data | At birth
  Proportion of HIV-infected women enrolled in antenatal care with a facility delivery
Maternal ART Adherence, evaluated using clinic registry data | At 3 and 6 months post ART initiation
  Proportion of expected ART medicines picked up at study clinics
Viral Suppression, evaluated using clinic registry data | Within 1 months of delivery
  Proportion of viral load samples with undetectable viral load (<20 copies/mL)
Mother-to-Child HIV Transmission Rate, evaluated using clinic registry data | 6 months postpartum
  Proportion of HIV-exposed infants testing positive for HIV

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Sherr, PhD, Principal Investigator — University of Washington
Locations (1):
- Manica Province, Chimoio, Manica Province, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
Patient- and aggregate facility-level data will be made available to users who request access to the data after a manuscript based on the primary study results is accepted for publication. User registration will be required in order to access or download files. As part of the registration process, users must agree to the conditions of use governing access to the public release data, including destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource. Registered users will receive user support, as well as information related to errors in the data, future releases, workshops, and publication lists. The information provided to users will not be used for commercial purposes, and will not be redistributed to third parties. Data from focus group discussions and key informant interviews will not be available because of human subjects protections constraints.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After a manuscript with primary study results is accepted for publication.
Access Criteria: User registration will be required in order to access or download files. As part of the registration process, users must agree to the conditions of use governing access to the public release data, including destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource. The information provided to users will not be used for commercial purposes, and will not be redistributed to third parties.

REFERENCES:
- [Background] Gimbel S, Voss J, Rustagi A, Mercer MA, Zierler B, Gloyd S, Coutinho Mde J, Cuembelo Mde F, Sherr K. What does high and low have to do with it? Performance classification to identify health system factors associated with effective prevention of mother-to-child transmission of HIV delivery in Mozambique. J Int AIDS Soc. 2014 Mar 24;17(1):18828. doi: 10.7448/IAS.17.1.18828. eCollection 2014. PMID 24666594
- [Background] Gimbel S, Rustagi AS, Robinson J, Kouyate S, Coutinho J, Nduati R, Pfeiffer J, Gloyd S, Sherr K, Granato SA, Kone A, Cruz E, Manuel JL, Zucule J, Napua M, Mbatia G, Wariua G, Maina M; with input from the SAIA study team. Evaluation of a Systems Analysis and Improvement Approach to Optimize Prevention of Mother-To-Child Transmission of HIV Using the Consolidated Framework for Implementation Research. J Acquir Immune Defic Syndr. 2016 Aug 1;72 Suppl 2(Suppl 2):S108-16. doi: 10.1097/QAI.0000000000001055. PMID 27355497
- [Background] Rustagi AS, Gimbel S, Nduati R, Cuembelo Mde F, Wasserheit JN, Farquhar C, Gloyd S, Sherr K; with input from the SAIA Study Team. Implementation and Operational Research: Impact of a Systems Engineering Intervention on PMTCT Service Delivery in Cote d'Ivoire, Kenya, Mozambique: A Cluster Randomized Trial. J Acquir Immune Defic Syndr. 2016 Jul 1;72(3):e68-76. doi: 10.1097/QAI.0000000000001023. PMID 27082507
- [Background] Gimbel S, Voss J, Mercer MA, Zierler B, Gloyd S, Coutinho Mde J, Floriano F, Cuembelo Mde F, Einberg J, Sherr K. The prevention of mother-to-child transmission of HIV cascade analysis tool: supporting health managers to improve facility-level service delivery. BMC Res Notes. 2014 Oct 21;7:743. doi: 10.1186/1756-0500-7-743. PMID 25335783
- [Background] Sherr K, Gimbel S, Rustagi A, Nduati R, Cuembelo F, Farquhar C, Wasserheit J, Gloyd S; With input from the SAIA Study Team. Systems analysis and improvement to optimize pMTCT (SAIA): a cluster randomized trial. Implement Sci. 2014 May 8;9:55. doi: 10.1186/1748-5908-9-55. PMID 24885976
- [Derived] Inguane C, Gimbel S, Soi C, Tavede E, Murgorgo F, Isidoro X, Sidat Y, Nassiaca R, Coutinho J, Cruz M, Agostinho M, Amaral F, Dinis A, Absjornsdottir K, Crocker J, Manaca N, Ramiro I, Pfeiffer J, de Fatima Cuembelo M, Sherr K. Assessing drivers of implementing "Scaling-up the Systems Analysis and Improvement Approach" for Prevention of Mother-to-Child HIV Transmission in Mozambique (SAIA-SCALE) over implementation waves. Implement Sci Commun. 2023 Jul 24;4(1):84. doi: 10.1186/s43058-023-00422-6. PMID 37488632
- [Derived] Sherr K, Asbjornsdottir K, Crocker J, Coutinho J, de Fatima Cuembelo M, Tavede E, Manaca N, Ronen K, Murgorgo F, Barnabas R, John-Stewart G, Holte S, Weiner BJ, Pfeiffer J, Gimbel S. Scaling-up the Systems Analysis and Improvement Approach for prevention of mother-to-child HIV transmission in Mozambique (SAIA-SCALE): a stepped-wedge cluster randomized trial. Implement Sci. 2019 Apr 27;14(1):41. doi: 10.1186/s13012-019-0889-z. PMID 31029171